CLINICAL TRIAL: NCT06872957
Title: Trapezius Muscle Activity During Wall-Slide Exercise: Natural Vs Corrected Head Posture
Brief Title: Trapezius Muscle Activities in the Natural Head Posture and Corrected Head Posture During Wall-Slide Exercise
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022 - 265
Record Dates: First submitted 2025-03-05; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Trapezius Muscle Atrophy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy individuals: Healthy individuals between the ages of 18 and 35 were included in the study. Activation of the upper trapezius, middle trapezius and lower trapezius were measured with 8-channel surface EMG Noraxon MiniDTS system (Noraxon, USA, Inc, Scottsdale, AZ), a non-invasive method measuring muscle activation, while the participants were performing wall-slide exercise with different head postures (natural head posture and corrected head posture)
  Interventions: Device: Surface Electromyography Noraxon MiniDTS system

INTERVENTIONS:
Device: Surface Electromyography Noraxon MiniDTS system — Trapezius muscle activities of 19 healthy individuals were measured with surface EMG Noraxon MiniDTS system (Noraxon, USA, Inc, Scottsdale, AZ) in the ascending, stationary and descending phases of the wall slide exercise under different head posture conditions: natural head posture and corrected head posture.

SUMMARY:
The goal of this observational study is to investigate the effect of head posture on trapezius muscle activity and ratios during wall slide exercise. The main question the study aims to answer is:

•How does the trapezius muscle activity change during wall slide exercise when performed with a natural head posture and the corrected head posture? The participants performed wall slide exercise with their natural head posture and the corrected posture. For both interventions, muscle activity of the lower, middle and upper trapezius was measured with surface electromyography(EMG) Noraxon MiniDTS system (Noraxon, USA, Inc, Scottsdale, AZ) in the ascending, stationary and descending phases of the exercise.

DETAILED DESCRIPTION:
Healthy individuals between the ages of 18 and 35 who have not had any pain in the upper extremity for the last 6 weeks, have musculoskeletal system pathologies of the upper extremity and/or any surgery were included in the study. Individuals who have had pain in the shoulder area for the last 6 weeks, had shoulder injury and/or shoulder surgery, have neurological, rheumatological or systemic diseases and body mass index (BMI) greater than 30 kg/m2 were excluded. Participants were asked to perform wall-slide exercise with both natural head posture and corrected head posture, separately. During the wall-slide exercise, muscle activations of upper trapezius (UT), middle trapezius (MT) and lower trapezius (LT) were measured with surface EMG Noraxon MiniDTS system (Noraxon, USA, Inc, Scottsdale, AZ) in the ascending, stationary and descending phases of the exercise.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals between the ages of 18 and 35
* Individuals who have not had any pain in the upper extremity for the last 6 weeks
* Individuals who do not have musculoskeletal system pathologies of the upper extremity and/or any surgery

Exclusion Criteria:

* Individuals who have had pain in the shoulder area for the last 6 weeks
* Individuals who had shoulder injury and/or shoulder surgery
* Individuals who have neurological, rheumatological or systemic diseases
* Individuals with body mass index (BMI) greater than 30 kg/m2

Ages: 18 Hours to 35 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy individuals between the ages of 18 and 35
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2022-03-05 (Actual); Study Completion 2022-03-05 (Actual)

PRIMARY OUTCOMES:
Trapezius muscle activity | Baseline
  Upper, middle and lower trapezius muscle activities were recorded through surface EMG.

CONTACTS AND LOCATIONS:
Overall Officials: Nihan Karataş, Prof., Principal Investigator — Gazi University
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Maenhout A, Benzoor M, Werin M, Cools A. Scapular muscle activity in a variety of plyometric exercises. J Electromyogr Kinesiol. 2016 Apr;27:39-45. doi: 10.1016/j.jelekin.2016.01.003. Epub 2016 Jan 28. PMID 26894494
- [Background] Kara D, Harput G, Duzgun I. Shoulder-Abduction Angle and Trapezius Muscle Activity During Scapular-Retraction Exercise. J Athl Train. 2021 Dec 1;56(12):1327-1333. doi: 10.4085/1062-6050-0053.21. PMID 34911072
- [Background] Cools AM, Dewitte V, Lanszweert F, Notebaert D, Roets A, Soetens B, Cagnie B, Witvrouw EE. Rehabilitation of scapular muscle balance: which exercises to prescribe? Am J Sports Med. 2007 Oct;35(10):1744-51. doi: 10.1177/0363546507303560. Epub 2007 Jul 2. PMID 17606671
- [Background] Cools AM, Declercq GA, Cambier DC, Mahieu NN, Witvrouw EE. Trapezius activity and intramuscular balance during isokinetic exercise in overhead athletes with impingement symptoms. Scand J Med Sci Sports. 2007 Feb;17(1):25-33. doi: 10.1111/j.1600-0838.2006.00570.x. Epub 2006 Jun 15. PMID 16774650
- [Background] Colado JC, Garcia-Masso X, Triplett NT, Calatayud J, Flandez J, Behm D, Rogers ME. Construct and concurrent validation of a new resistance intensity scale for exercise with thera-band(R) elastic bands. J Sports Sci Med. 2014 Dec 1;13(4):758-66. eCollection 2014 Dec. PMID 25435767